CLINICAL TRIAL: NCT00673101
Title: Evaluation of Liver Fibrosis Using FibroScan and Non-invasive Biochemical Markers in Patients Treated With Methotrexate
Brief Title: Prospective Evaluation of FibroScan in Patients Treated With Methotrexate
Acronym: Methoscan
Status: Completed | Type: Observational
Sponsor: Association HGE CHU Bordeaux Sud (Other)
Responsible Party: Principal Investigator, de Ledinghen, Professor, Association HGE CHU Bordeaux Sud
Other Study IDs: 05-07
Record Dates: First submitted 2008-05-06; First posted 2008-05-07 (Estimated); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Liver Fibrosis
Keywords: liver fibrosis, cirrhosis; FibroScan; transient elastography; elastometry; methotrexate; non invasive blood markers; FibroTest; treatment
MeSH Terms: conditions — Liver Cirrhosis; Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of this study is to evaluate liver fibrosis using FibroScan and biochemical markers in patients treated with methotrexate.

DETAILED DESCRIPTION:
Methotrexate (MTX) is an effective treatment for induction of remission and maintenance in patients with Crohn's disease, rheumatoid arthritis, or psoriasis which may induce liver fibrosis with high cumulative doses. Transient elastography (FibroScan) is a new non-invasive rapid, reproducible and bed-side method, allowing assessment of liver fibrosis by measurement of liver stiffness. A preliminary study (Laharie et al, Alimentary Pharmaceutical Therapeutics 2006) had shown that significant liver fibrosis was rare in Crohn's disease patients treated with a high dose of methotrexate. FibroScan was a reliable non-invasive method to detect liver fibrosis which could be recommended in these patients. Therefore, liver biopsy could be performed only with patients with high FibroScan values and/or with chronic liver enzymes abnormalities. However, further longitudinal and prospective studies are mandatory to confirm these preliminary data, in patients with crohn's disease but also with rheumatoid arthritis and psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects, ≥18 years of age.
* Patient treated with Methotrexate.
* Written informed consent

Exclusion Criteria:

* Patients refusing to participate to the study and to provide written informed consent
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated by Methotrexate
Sampling Method: Non-Probability Sample
Enrollment: 1871 (Actual)
Dates: Start 2006-01; Primary Completion 2019-07 (Actual); Study Completion 2019-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thierry Schaeverbeke, MD, PhD, Principal Investigator — University Hospital, Bordeaux; Edouard Chabrun, MD, Principal Investigator — Gastroenterology and Hepatology Unit, Haut-Lévêque Hospital, 33604 Pessac, France; Thomas Hubiche, MD, Principal Investigator — University Hospital, Bordeaux; Marie-Sylvie Doutre, MD, PhD, Principal Investigator — University Hospital, Bordeaux; Maïté Longy-Boursier, MD, PhD, Principal Investigator — CHU de Bodeaux; Jean-Luc Pellegrin, MD, PhD, Principal Investigator — University Hospital, Bordeaux; Juliette Foucher, MD, Principal Investigator — Gastroenterology and Hepatology Unit, Haut-Lévêque Hospital, 33604 Pessac, France; Franck Zerbib, MD PhD, Principal Investigator — Gastroenterology and Hepatology Unit, Saint-André Hospital, 33075 Bordeaux, Cedex, France; David Laharie, MD PhD, Study Director — University Hospital, Bordeaux
Locations (1):
- Hopital du Haut Leveque, Pessac, France